CLINICAL TRIAL: NCT01345253
Title: GSK1550188 A 52 Week Study of Belimumab Versus Placebo in the Treatment of Subjects With Systemic Lupus Erythematosus (SLE) Located in Northeast Asia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113750
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Results first posted 2016-12-02 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLEDAI; Asia; placebo; BLys; PGA; BILAG; systemic lupus erythematosus; SELENA; Lupus; SRI; efficacy; B cell; SLE Flare Index; belimumab; safety; phase III; B lymphocyte
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Belimumab (Experimental): 10mg/kg
  Interventions: Drug: Belimumab
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Belimumab — 10mg/kg administered intravenously. Dosing at Weeks 0, 2, and 4, then every 4 weeks through Week 48, with a final evaluation at Week 52. All study subjects will receive standard SLE therapies during the study.
  Arms: Belimumab
Drug: Placebo — Administered intravenously. Dosing at Weeks 0, 2, and 4, and then every 4 weeks through Week 48, with a final evaluation at Week 52. All study subjects will receive standard SLE therapies during the study.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of belimumab in addition to standard therapy compared to placebo in subjects in Northeast Asia with systemic lupus erythematosus (SLE) over a 52 week period.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the efficacy and safety of belimumab 10mg/kg administered intravenously (IV) every 4 weeks compared to placebo, in patients with SLE when added to standard of care therapy, as measured by the SLE Responder Index (SRI) at 52 weeks, defined by a composite endpoint using SELENA SLEDAI score, Physician's Global Assessment (PGA) and BILAG A and B organ domain scores.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older.
* Have a clinical diagnosis of SLE according to the American College of Rheumatology (ACR) classification criteria.
* Have active SLE disease.
* Have positive anti-nuclear antibody (ANA) test results.
* Are on a stable SLE treatment regimen.
* Females of childbearing age are willing to use appropriate contraception

Exclusion Criteria:

* Have received treatment with any B cell targeted therapy at any time.
* Have received a biologic investigational agent in the past year.
* Have received 3 or more courses of systemic corticosteroids in the past year.
* Have received intravenous (IV) cyclophosphamide within 180 days prior to Day 0.
* Have severe lupus kidney disease.
* Have active central nervous system (CNS) lupus.
* Have had a major organ transplant.
* Have significant unstable or uncontrolled acute or chronic diseases or conditions not due to SLE.
* Have a planned surgical procedure.
* Cancer within the last 5 years, except for adequately treated skin cancer, or carcinoma in situ of the uterine cervix.
* Have required management of acute or chronic infections in the past 60 days.
* Have current drug or alcohol abuse or dependence.
* Have a historically positive test, or test positive at screening for HIV, Hepatitis B, or Hepatitis C.
* Have an IgA deficiency.
* Have severe laboratory Abnormalities.
* Have had anaphylactic reaction to X-ray contrast agents or biologic agents.
* Suicidal behavior or ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2011-05-23 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2018-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (32):
- China (15):
  - GSK Investigational Site, Hefei, Anhui
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Harbin, Heilongjiang
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Suzhou, Jiangsu
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Kunming, Yunnan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
- Japan (12):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
- South Korea (5):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do

REFERENCES:
- [Background] Zhang F, Bae SC, Bass D, Chu M, Egginton S, Gordon D, Roth DA, Zheng J, Tanaka Y. A pivotal phase III, randomised, placebo-controlled study of belimumab in patients with systemic lupus erythematosus located in China, Japan and South Korea. Ann Rheum Dis. 2018 Mar;77(3):355-363. doi: 10.1136/annrheumdis-2017-211631. Epub 2018 Jan 2. PMID 29295825
- [Derived] Nikolopoulos D, Cetrez N, Lindblom J, Parodis I. Neuropsychiatric involvement in systemic lupus erythematosus contributes to organ damage beyond the nervous system: a post-hoc analysis of 5 phase III randomized clinical trials. Rheumatol Int. 2024 Sep;44(9):1679-1689. doi: 10.1007/s00296-024-05667-5. Epub 2024 Aug 8. PMID 39115551
- [Derived] Jagerback S, Gomez A, Parodis I. Predictors of renal flares in systemic lupus erythematosus: a post-hoc analysis of four phase III clinical trials of belimumab. Rheumatology (Oxford). 2025 Feb 1;64(2):623-631. doi: 10.1093/rheumatology/keae023. PMID 38216728
- [Derived] Suh CH, Lee Y, Yoo SB, Quasny H, Navarro Rojas AA, Hammer A, Song YW, Kang YM, Cho CS, Park W, Kwok SK, Lee SG, Chung WT, Bae SC. Efficacy and safety of intravenous belimumab in a subgroup of South Korean patients with systemic lupus erythematosus enrolled into a Phase 3, randomized, placebo-controlled trial in North East Asia. Int J Rheum Dis. 2024 Jan;27(1):e14997. doi: 10.1111/1756-185X.14997. Epub 2023 Dec 23. PMID 38140854
- [Derived] Gomez A, Jagerback S, Sjowall C, Parodis I. Belimumab and antimalarials combined against renal flares in patients treated for extra-renal systemic lupus erythematosus: results from 4 phase III clinical trials. Rheumatology (Oxford). 2024 Feb 1;63(2):338-348. doi: 10.1093/rheumatology/kead253. PMID 37228028
- [Derived] Zhang F, Zheng J, Li Y, Wang G, Wang M, Su Y, Gu J, Li X, Bass D, Chu M, Curtis P, DeRose K, Kurrasch R, Lowe J, Meizlik P, Roth DA. Phase 3, long-term, open-label extension period of safety and efficacy of belimumab in patients with systemic lupus erythematosus in China, for up to 6 years. RMD Open. 2022 Apr;8(1):e001669. doi: 10.1136/rmdopen-2021-001669. PMID 35428697
- [Derived] Gupta SV, Fanget MC, MacLauchlin C, Clausen VA, Li J, Cloutier D, Shen L, Robbie GJ, Mogalian E. Clinical and Preclinical Single-Dose Pharmacokinetics of VIR-2218, an RNAi Therapeutic Targeting HBV Infection. Drugs R D. 2021 Dec;21(4):455-465. doi: 10.1007/s40268-021-00369-w. Epub 2021 Nov 6. PMID 34741731
- [Derived] Zhou X, Lee TI, Zhu M, Ma P. Prediction of Belimumab Pharmacokinetics in Chinese Pediatric Patients with Systemic Lupus Erythematosus. Drugs R D. 2021 Dec;21(4):407-417. doi: 10.1007/s40268-021-00363-2. Epub 2021 Oct 9. PMID 34628605
- [Derived] Brunner HI, Abud-Mendoza C, Mori M, Pilkington CA, Syed R, Takei S, Viola DO, Furie RA, Navarra S, Zhang F, Bass DL, Eriksson G, Hammer AE, Ji BN, Okily M, Roth DA, Quasny H, Ruperto N. Efficacy and safety of belimumab in paediatric and adult patients with systemic lupus erythematosus: an across-study comparison. RMD Open. 2021 Sep;7(3):e001747. doi: 10.1136/rmdopen-2021-001747. PMID 34531304
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of a 52 week blinded treatment period in Northeast Asia (China, Japan, Korea) which was followed by an optional open-label (OL) extension period in China for evaluation of belimumab in participants (par.) with active systemic lupus erythematosus (SLE).
Pre-assignment Details: A total of 707 par. were randomized, 705 received at least 1 dose of investigational product (Safety Population), 677 par. were included in the primary efficacy population (MITT Population) of which 663 were evaluable for the primary endpoint. The participant flow and baseline characteristics are presented for MITT Population (Pop).
Groups:
- Placebo: Participants received placebo intravenously (IV) on Day 0, Day 14, Day 28 and then every 28 days until Week 48 of the double-blind period. All China participants who completed double-blind period and eligible to enter open-label phase received belimumab 10 milligrams (mg)/kilogram (kg) up to Year 5 Week 28.
- Belimumab 10 mg/kg: Participants received belimumab 10 mg/kg IV on Day 0, Day 14, Day 28 and then every 28 days until Week 48 of the double-blind period. All China participants who completed double-blind period and eligible to enter open-label phase received belimumab 10 mg/kg up to Year 5 Week 28.
Period: Double-blind (DB) Phase (52 Weeks)
Arm/Group | Placebo | Belimumab 10 mg/kg
Started | 226 | 451
Completed | 170 | 372
Not Completed | 56 | 79
Not completed — Adverse Event | 22 | 27
Not completed — Lack of Efficacy | 11 | 7
Not completed — Protocol Violation | 1 | 5
Not completed — Met Protocol Defined Stopping Criteria | 6 | 1
Not completed — Lost to Follow-up | 3 | 8
Not completed — Physician Decision | 4 | 12
Not completed — Withdrawal by Subject | 9 | 19
Period: Open-label Phase (Up to Year 5 Week 44)
Arm/Group | Placebo | Belimumab 10 mg/kg
Started | 134 (Only eligible China par. enrolled in OL phase from MITT + additional 9 China par. from Safety Pop) | 290 (Only eligible China par. enrolled in OL phase from MITT + additional 16 China par. from Safety Pop)
Completed | 69 | 146
Not Completed | 65 | 144
Not completed — Adverse Event | 7 | 18
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 3 | 7
Not completed — Protocol Violation | 2 | 5
Not completed — Lost to Follow-up | 4 | 6
Not completed — Physician Decision | 11 | 24
Not completed — Withdrawal by Subject | 37 | 82
Not completed — Not Recorded | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Belimumab 10 mg/kg | Total
Number analyzed (Participants) | 226 | 451 | 677
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.7 (9.18) | 32.3 (9.65) | 32.1 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 419 | 629
  Male | 16 | 32 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central/South Asian Heritage | 2 | 4 | 6
  Asian - East Asian Heritage | 195 | 403 | 598
  Asian - Japanese Heritage | 24 | 40 | 64
  Asian - South East Asian Heritage | 4 | 3 | 7
  Asian - Mixed Race | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Achieving Systemic Lupus Erythematosus (SLE) Responder Index (SRI) Response Rate at Week 52 for Double-blind Phase.
Description: SRI response is a composite index, defined as the percent of participants with >=4 point reduction from Baseline in safety of estrogen in lupus national assessment (SELENA) systemic lupus erythematosus disease activity index (SLEDAI) score and no worsening (increase of < 0.30 points from Baseline) in physicians global assessment (PGA) and no new British isles lupus assessment group (BILAG) A organ domain score or 2 new BILAG B organ domain scores compared with Baseline at the time of assessment (at Week 52 of the blinded period). A SELENA SLEDAI score of 0 would suggest no lupus activity; while a score of 105 is the maximum calculable if all items were scored as being present from active lupus. PGA ranges from 0 (no activity) to 3 (severe activity). BILAG has no range. The higher thresholds of SELENA SLEDAI improvement (i.e., SRI5, SRI6, and SRI7) indicates a higher response (SRI5 is a 5 point SELENA SLEDAI reduction, SRI6 is a 6 point reduction, and SRI7 is a 7 point reduction).
Time Frame: Week 52
Population: Modified Intention-to-Treat (MITT) Population: all participants who were randomized and treated with at least one dose of study treatment, with exclusion of participants from the site 086485.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 217 | 446
Percentage of participants | 40.1 | 53.8
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.99, 95% CI 2-sided [1.40 to 2.82] — Odds Ratio (95% CI) and p-value were estimated by a logistic regression model with independent variables treatment group, country, Baseline SELENA SLEDAI score (<=9 vs. >=10) and complement (C) levels (low C3 and/or C4 vs. no low C3 or C4)

2. Secondary Outcome: Percent of Participants With >=4 Point Reduction From Baseline in SELENA SLEDAI Score at Week 52 for Double-blind Phase.
Description: The SELENA SLEDAI score is a weighted index for assessing SLE disease activity in which signs and symptoms, laboratory tests and physician's assessment for each of 9 organ system were given a weighted score and summed if present at the time of the visit or in the preceding 10 days. A SELENA SLEDAI score of 0 would suggest no lupus activity; while a score of 105 is the maximum calculable if all items were scored as being present from active lupus. A decrease of 4 points or more equates to a clinically meaningful improvement. The Baseline value of a variable is defined as the value of the variable measured at Day 0 prior to dosing. In case of multiple results on Day 0 prior to dosing, the latest result was used. If a Day 0 value was not available, the last available value prior to Day 0 was used.
Time Frame: Baseline (Day 0) and Week 52
Population: MITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 218 | 447
Percentage of participants | 42.2 | 55.7
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.00, 95% CI 2-sided [1.41 to 2.83] — Odds Ratio (95% CI) and p-value were estimated by a logistic regression model with independent variables treatment group, country, Baseline SELENA SLEDAI score (<=9 vs. >=10) and complement levels (low C3 and/or C4 vs. no low C3 or C4)

3. Secondary Outcome: Percent of Participants With SRI7 Response at Week 52 for Double-blind Phase.
Description: SRI7 response is defined as the percent of participants with >=7 point reduction from Baseline in SELENA SLEDAI score and no worsening (increase of < 0.30 points from Baseline) in PGA and no new BILAG A organ domain score or 2 new BILAG B organ domain scores compared with Baseline at the time of assessment (at Week 52 of the blinded period). A SELENA SLEDAI score of 0 would suggest no lupus activity; while a score of 105 is the maximum calculable if all items were scored as being present from active lupus. PGA ranges from 0 (no activity) to 3 (severe activity). BILAG has no range. The higher thresholds of SELENA SLEDAI improvement (i.e., SRI5, SRI6, and SRI7) indicates a higher response (SRI5 is a 5 point SELENA SLEDAI reduction, SRI6 is a 6 point reduction, and SRI7 is a 7 point reduction).
Time Frame: Baseline (Day 0) and Week 52
Population: MITT Population. Only those participants available at the specified time point were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 183 | 367
Percentage of participants | 23.5 | 32.4
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.0116, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.13 to 2.74] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Days of Daily Prednisone Dose <=7.5 mg/Day and/or Reduced by 50 Percent From Baseline Over 52 Weeks for Double-blind Phase.
Description: Number of days of daily prednisone dose <=7.5 mg/day and/or reduced by 50 percent over time through each scheduled visit during the blinded period were compared between belimumab and placebo using Rank ANCOVA model which was used for comparing belimumab and placebo. The independent variables in the model included treatment group, Baseline prednisone dose level, country, Baseline SELENA SLEDAI score (<=9 vs. >=10) and complement levels (low C3 and/or C4 vs. no low C3 or C4). This analysis was perfomed on the participants who used prednisone >7.5 mg/day at Baseline.
Time Frame: Week 52
Population: MITT Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 184 | 352
Days | 0.0 [0.0 to 172.0] | 0.0 [0.0 to 213.5]
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.0288, Rank ANCOVA

5. Secondary Outcome: Time to First Severe SLE Flare Index (SFI) Flare Over 52 Weeks for Double-blind Phase.
Description: Time to first severe SLE flare is defined as the number of days from first treatment until the participant had an event (event date-treatement start date +1). If a participant had a severe SFI flare and received protocol restricted medication then the event date was the earliest of the first severe SFI flare date, and the treatment failure date. Analysis of severe SFI flare was performed on the modified SELENA SLEDAI SLE flare index in which the modification excluded severe flares that were triggered only by an increase in SELENA SLEDAI score to >12. Analysis was from Cox proportional hazards model for the comparison between belimumab and placebo adjusting for country, Baseline SELENA SLEDAI score (<=9 vs. >=10) and complement levels (low C3 and/or C4 vs. no low C3 or C4).
Time Frame: 52 weeks
Population: MITT Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 226 | 451
Days | NA [NA to NA] — Due to low event rates of participants in both treatment groups having severe SFI flares, the median time and interquartile range could not be estimated. | NA [NA to NA] — Due to low event rates of participants in both treatment groups having severe SFI flares, the median time and interquartile range could not be estimated.
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.0004, Regression, Cox; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.34 to 0.73]

6. Secondary Outcome: Percent of Participants Achieving SLE SRI Response Rate for Open-label (OL) Phase
Description: SRI response is a composite index, defined as the percent of participants with >=4 point reduction from Baseline in SELENA SLEDAI score and no worsening (increase of < 0.30 points from Baseline) in PGA and no new BILAG A organ domain score or 2 new BILAG B organ domain scores compared with Baseline at time of assessment. Excludes participants with a SELENA SLEDAI score <4 at baseline. Participants randomized to belimumab in double-blinded (DB) phase, Baseline is last available value before first belimumab dose received in DB phase. Participants randomized to placebo in DB phase, Baseline is last available value before receiving first belimumab dose in OL phase. Observed case data are presented.Year 6 Week 48 is the Exit Visit obtained by slotting the Exit Visit to Week 48. A SELENA SLEDAI score of 0 (no lupus activity) and a score of 105 (maximum). PGA ranges from 0 (no activity) to 3 (severe activity). BILAG has no range.
Time Frame: Weeks 24 and 48 for Years 2, 3, 4, 5 and 6
Population: Efficacy Population: all participants in China who received at least 1 dose of belimumab during open-label phase, exclusive of site 086485. Only those participants available at the specified time points were analyzed (represented by n=x).
Measure: Number; unit: Percentage of participants
Groups:
- Belimumab 10mg/kg (Open-label Phase): All eligible China participants who had received placebo and belimumab in DB period and entered open-label phase to receive belimumab 10 mg/kg over 1 hour every 28 days from first belimumab date through end of open-label phase.
Arm/Group | Belimumab 10mg/kg (Open-label Phase)
Number analyzed (Participants) | 399
Percentage of participants
  Week 24, Year 2, n=326: number analyzed (Participants) | 326
  Week 24, Year 2, n=326 | 66.0
  Week 48, Year 2, n=299: number analyzed (Participants) | 299
  Week 48, Year 2, n=299 | 69.6
  Week 24, Year 3, n=271: number analyzed (Participants) | 271
  Week 24, Year 3, n=271 | 72.3
  Week 48, Year 3, n=247: number analyzed (Participants) | 247
  Week 48, Year 3, n=247 | 70.9
  Week 24, Year 4, n=233: number analyzed (Participants) | 233
  Week 24, Year 4, n=233 | 71.7
  Week 48, Year 4, n=194: number analyzed (Participants) | 194
  Week 48, Year 4, n=194 | 76.8
  Week 24, Year 5, n= 156: number analyzed (Participants) | 156
  Week 24, Year 5, n= 156 | 81.4
  Week 48, Year 5, n= 82: number analyzed (Participants) | 82
  Week 48, Year 5, n= 82 | 80.5
  Week 24, Year 6, n= 36: number analyzed (Participants) | 36
  Week 24, Year 6, n= 36 | 86.1
  Week 48, Year 6, n= 5: number analyzed (Participants) | 5
  Week 48, Year 6, n= 5 | 60.0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-SAEs were collected from study treatment start and until 16 weeks after the last infusion. The data presented for belimumab open-label group represents safety events period starting from the first belimumab date and up to Year 6 Week 44.
Description: SAEs and non-serious AEs were reported for the Safety Population consisted of all participants who received at least one dose of study drug. The first belimumab date was first dose received in DB phase for participants randomized to belimumab in DB phase; first dose received in OL phase for participants randomized to placebo in DB phase.
Groups:
- Placebo (Double-blind Phase): Participants received placebo intravenously (IV) on Day 0, Day 14, Day 28 and then every 28 days until Week 48 of the blinded period.
- Belimumab 10 mg/kg (Double-blind Phase): Participants received belimumab 10 miligrams (mg)/kilogram (kg) IV on Day 0, Day 14, Day 28 and then every 28 days until Week 48 of the blinded period.
- Belimumab 10 mg/kg (Open-label Phase): All eligible China participants who had received placebo and belimumab in DB period and entered open-label phase to receive belimumab 10 mg/kg over 1 hour every 28 days from first belimumab date through end of open-label phase.
Arm/Group | Placebo (Double-blind Phase) | Belimumab 10 mg/kg (Double-blind Phase) | Belimumab 10 mg/kg (Open-label Phase)
All-Cause Mortality (participants affected / at risk) | 1/235 | 0/470 | 1/424
Serious Adverse Events (participants affected / at risk) | 43/235 | 58/470 | 96/424
Other Adverse Events (participants affected / at risk) | 108/235 | 207/470 | 263/424
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind Phase) (N=235) | Belimumab 10 mg/kg (Double-blind Phase) (N=470) | Belimumab 10 mg/kg (Open-label Phase) (N=424)
Herpes zoster (Infections and infestations) | 2 | 6 | 6
Pneumonia (Infections and infestations) | 1 | 2 | 4
Appendicitis (Infections and infestations) | 0 | 2 | 2
Lung infection (Infections and infestations) | 2 | 0 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 2 | 0
Salmonella sepsis (Infections and infestations) | 2 | 0 | 0
Skin infection (Infections and infestations) | 1 | 1 | 0
Arthritis salmonella (Infections and infestations) | 0 | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cellulitis streptococcal (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastrointestinal fungal infection (Infections and infestations) | 1 | 0 | 0
Infectious colitis (Infections and infestations) | 0 | 1 | 0
Lymph node tuberculosis (Infections and infestations) | 1 | 0 | 0
Meningitis tuberculous (Infections and infestations) | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Spleen tuberculosis (Infections and infestations) | 1 | 0 | 0
Tuberculosis liver (Infections and infestations) | 1 | 0 | 0
Tuberculous pleurisy (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Lupus nephritis (Renal and urinary disorders) | 5 | 5 | 12
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1
Lupus cystitis (Renal and urinary disorders) | 0 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Pyrexia (General disorders) | 4 | 2 | 1
Generalised oedema (General disorders) | 1 | 0 | 0
Polyserositis (General disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1
Allergic colitis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Lupus pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lupus encephalitis (Nervous system disorders) | 1 | 1 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Arterial rupture (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Lupus vasculitis (Vascular disorders) | 0 | 1 | 0
Necrosis ischaemic (Vascular disorders) | 0 | 1 | 2
Phlebitis (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0
SLE arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lupus pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lupus pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 1
Periorbital infection (Infections and infestations) | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 1
Ludwig angina (Infections and infestations) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 1
Cutaneous tuberculosis (Infections and infestations) | 0 | 0 | 1
Breast abscess (Infections and infestations) | 0 | 0 | 1
Bartholin's abscess (Infections and infestations) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Benign ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Neuropsychiatric lupus (Nervous system disorders) | 0 | 0 | 1
Noninfectious myelitis (Nervous system disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Granuloma (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 1
Endometrial thickening (Reproductive system and breast disorders) | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Protein urine present (Investigations) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind Phase) (N=235) | Belimumab 10 mg/kg (Double-blind Phase) (N=470) | Belimumab 10 mg/kg (Open-label Phase) (N=424)
Upper respiratory tract infection (Infections and infestations) | 39 | 65 | 149
Nasopharyngitis (Infections and infestations) | 26 | 56 | 24
Viral upper respiratory tract infection (Infections and infestations) | 15 | 33 | 59
Upper respiratory tract infection bacterial (Infections and infestations) | 12 | 16 | 37
Diarrhoea (Gastrointestinal disorders) | 14 | 28 | 28
Pyrexia (General disorders) | 17 | 28 | 36
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 30 | 30
Headache (Nervous system disorders) | 16 | 23 | 20
Urinary tract infection (Infections and infestations) | 11 | 21 | 41
Herpes zoster (Infections and infestations) | 10 | 23 | 34
Urinary tract infection bacterial (Infections and infestations) | 2 | 20 | 23
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 11 | 24

LIMITATIONS AND CAVEATS:
The primary objective for DB was efficacy and the participant flow is aligned with the MITT population. The primary objective for OL is safety and includes only China par. from DB + additional 25 China par. from the Safety Pop who were not in MITT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.